CLINICAL TRIAL: NCT03614494
Title: Piroxicam and Levonorgestrel Co-treatment for Emergency Contraception: Randomised Controlled Trial
Brief Title: Piroxicam and Levonorgestrel Co-treatment for Emergency Contraception
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. Hang Wun Raymond Li (Other)
Collaborators: The Family Planning Association of Hong Kong (Other)
Responsible Party: Sponsor-Investigator, Dr. Hang Wun Raymond Li, Clinical Associate Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW18-003
Record Dates: First submitted 2018-07-29; First posted 2018-08-03 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2023-11

CONDITIONS: Emergency Contraception
Keywords: Piroxicam; Levonorgestrel; Placebo; Randomised controlled control; Emergency contraception
MeSH Terms: interventions — Piroxicam; Levonorgestrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piroxicam (Active Comparator): Piroxicam 40 mg (in 2 tablets) + levonorgestrel 1.5 mg single oral dose
  Interventions: Drug: Piroxicam 40 mg; Drug: Levonorgestrel 1.5mg
- Placebo (Placebo Comparator): Placebo (2 tablets) + levonorgestrel 1.5 mg single oral dose
  Interventions: Drug: Levonorgestrel 1.5mg

INTERVENTIONS:
Drug: Piroxicam 40 mg — Additional co-treatment
  Arms: Piroxicam
Drug: Levonorgestrel 1.5mg — Standard treatment

SUMMARY:
This is a randomised controlled trial aimed at comparing the efficacy of levonorgestrel (LNG) co-administered with piroxicam or placebo for oral emergency contraception (EC). Piroxicam is a non-steroidal anti-inflammatory drug (NSAID) commonly used as a pain-killer in inflammatory conditions. Efficacy will be measured as the percentage of pregnancies prevented.

DETAILED DESCRIPTION:
Objective: To compare the percentage of pregnancies prevented by LNG co-administered with piroxicam or placebo for oral emergency contraception (EC) by a randomised controlled trial.

Hypothesis to be tested: LNG plus piroxicam has higher percentage of pregnancies prevented compared with LNG plus placebo for oral emergency contraception.

Design and subjects: This will be a prospective, randomised placebo-controlled clinical trial. Women attending the Family Planning Association of Hong Kong for oral EC within 72 hours of unprotected sexual intercourse will be recruited.

Study instruments: Prospective follow-up of subjects in the clinic for the primary and secondary outcomes.

Interventions: Eligible subjects will be randomised to receive one of the two treatment regimens, i.e. Group A: a single dose of LNG 1.5 mg and piroxicam 40 mg, or Group B: a single dose of LNG 1.5mg and placebo under direct supervision.

Main outcome measures: Percentage of pregnancies prevented (PPP) is the primary outcome measure. Secondary outcome measures include failure rate, rate of occurrence of side effects and pattern of the menstruation following EC.

Data analysis:The percentage of pregnancies prevented, failure rate and rate of occurrence of side effects will be compared between groups using Fisher-Exact test. Continuous variables regarding menstrual pattern between the two groups will be compared by Mann-Whitney U test.

Expected results: LNG plus piroxicam has a higher PPP compared to LNG plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* healthy women aged 18 years or above;
* requesting emergency contraception within 72 h of a single act of unprotected intercourse in the current menstrual cycle;
* having menstrual cycles between 24 and 42 days
* willing to abstain from further acts of unprotected intercourse and;
* available for follow-up over the next 6 weeks.

Exclusion Criteria:

* post-abortion or postpartum and period have not yet returned,
* being on prescription drugs currently
* having unprotected intercourse in this cycle more than 72 hours or more than once before attending the clinic,
* being found pregnant at the time of presentation,
* breastfeeding,
* having been sterilized (or partner having been sterilized) or having intrauterine contraceptive device in-situ,
* uncertain about the date of the last menstrual period,
* having used hormonal contraceptive (including EC pill) or NSAID in the current or past one cycle,
* having history of asthma, urticarial or other allergic reactions to piroxicam, aspirin or other NSAIDs,
* having history of ischaemic heart disease in the past one year
* having history of pelvic ulcer disease and/or gastrointestinal bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females are eligible
Enrollment: 860 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hang Wun Raymond Li, MD, FRCOG, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - The Family Planning Association of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
To be assessed and endorsed by the investigation team based on the exact study protocol suggested by the other researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication of results
Access Criteria: To be assessed and endorsed by the investigation team based on the exact study protocol suggested by the other researchers.

REFERENCES:
- [Derived] Li RHW, Lo SST, Gemzell-Danielsson K, Fong CHY, Ho PC, Ng EHY. Oral emergency contraception with levonorgestrel plus piroxicam: a randomised double-blind placebo-controlled trial. Lancet. 2023 Sep 9;402(10405):851-858. doi: 10.1016/S0140-6736(23)01240-0. Epub 2023 Aug 16. PMID 37597523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 860 women were recruited, all following the recruitment criteria, at the Family Planning Association of Hong Kong, between 20 August 2018 and 30 August 2022.
Pre-assignment Details: No per-assignment drop-out.
Groups:
- Piroxicam: Piroxicam 40 mg (in 2 tablets) + levonorgestrel 1.5 mg single oral dose
  430 women enrolled and received study drugs as per protocol. 12 lost to follow-up. 418 women who were efficacy-evaluable.
- Placebo: Placebo (2 tablets) + levonorgestrel 1.5 mg single oral dose
  430 women enrolled and received study drugs as per protocol. 12 lost to follow-up. 418 women who were efficacy-evaluable.
Period: Overall Study
Arm/Group | Piroxicam | Placebo
Started | 430 | 430
Completed | 418 | 418
Not Completed | 12 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Piroxicam | Placebo | Total
Number analyzed (Participants) | 430 | 430 | 860
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 430 | 430 | 860
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (5.9) | 31.9 (5.8) | 32.2 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 430 | 430 | 860
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 416 | 417 | 833
  Other Asians | 5 | 8 | 13
  Caucasian | 8 | 4 | 12
  African | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Hong Kong | 430 | 430 | 860
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 21.7 (3.3) | 21.9 (3.4) | 21.8 (3.3)
Coitus-treatment interval [Mean (Standard Deviation); unit: hours] | 23.6 (15.2) | 24.4 (15.7) | 24.0 (15.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Pregnancies Prevented
Description: (number of expected pregnancies - number of observed pregnancies) / number of expected pregnancies. The number of expected pregnancies is calculated based on the cycle day on which unprotected sexual intercourse occurred in each woman according to the model published by Trussel et al (Trussell J et al, Contraception 2003; 67:259-265).
Time Frame: 1 month
Population: efficacy-evaluable participants
Measure: Number; unit: percentage of pregnancies prevented
Arm/Group | Piroxicam | Placebo
Number analyzed (Participants) | 418 | 418
percentage of pregnancies prevented | 94.7 | 63.3
Statistical Analysis 1: Comparison: Piroxicam vs Placebo; Test type: Superiority; p < 0.0001, Chi-squared; Risk Difference (RD) = 31.4, 95% CI 2-sided [26.2 to 36.4]

2. Secondary Outcome: Pregnancy Rate
Description: number of participants who were pregnant / number of efficacy-evaluable participants
Time Frame: 1 month
Population: Participants who completed follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Piroxicam | Placebo
Number analyzed (Participants) | 418 | 418
Participants | 1 | 7
Statistical Analysis 1: Comparison: Piroxicam vs Placebo; Test type: Superiority; p = 0.036, Logistic regression, Firth's bias reduct; Odds Ratio (OR) = 0.197, 95% CI 2-sided [0.021 to 0.906]

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Piroxicam | Placebo
All-Cause Mortality (participants affected / at risk) | 0/430 | 0/430
Serious Adverse Events (participants affected / at risk) | 0/430 | 0/430
Other Adverse Events (participants affected / at risk) | 117/418 | 133/418
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Piroxicam (N=418) | Placebo (N=418)
Nausea (Gastrointestinal disorders) | 32 | 34
Fatigue / weakness (General disorders) | 43 | 52
Dizziness (Nervous system disorders) | 26 | 26
Headache (Nervous system disorders) | 21 | 27
Breast tenderness (Reproductive system and breast disorders) | 25 | 23
Lower abdominal pain (Gastrointestinal disorders) | 31 | 29
Stomachache (Gastrointestinal disorders) | 12 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT03614494/Prot_SAP_000.pdf